CLINICAL TRIAL: NCT01080820
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Study of the Safety, Tolerability and Pharmacokinetics of CMX157 in Healthy Adult Volunteers.
Brief Title: A Safety, Tolerability and Pharmacokinetic Study of a Single Dose of CMX157 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Margaret Anderson, Clinical Development Manager, Chimerix, Inc
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CMX157-101/A01
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Last update posted 2011-07-04 (Estimated); Status verified 2011-06

CONDITIONS: Healthy
Keywords: Healthy adult volunteers; Pharmacokinetics
MeSH Terms: interventions — hexadecyloxypropyl 9-(2-(phosphonomethoxy)propyl)adenine; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo + Viread (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Viread
- Viread (Active Comparator)
  Interventions: Drug: Viread
- CMX157 + Viread (Experimental)
  Interventions: Drug: CMX157; Drug: Viread

INTERVENTIONS:
Drug: CMX157 — One single oral dose of CMX157 will be administered and the option of receiving a single dose of 300mg Viread will be offered 4-8 weeks after the CMX157 dose.
  Arms: CMX157 + Viread
Drug: Placebo — One single oral dose of placebo will be administered and the option of receiving a single dose of 300mg Viread will be offered 4-8 weeks after the placebo dose.
  Arms: Placebo + Viread
Drug: Viread — One single oral dose of 300mg Viread.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of CMX157 and the amount of CMX157 that reaches the blood stream, the manner in which the body processes CMX157 and the time that it takes to eliminate CMX157 following one oral dose when given to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of non-childbearing potential, 18 to 55 years of age. Males must be able and willing to use adequate contraceptive methods throughout the study.

Exclusion Criteria:

1. Currently nursing females, pregnant females, or females of child-bearing potential.
2. Hypersensitivity to tenofovir.
3. Use of any antiviral, corticosteroid, immunosuppressive, or anticoagulant prescription drug within 4 weeks prior to enrollment. Use of any other prescription drug within 14 days prior to enrollment.
4. Use of any over-the-counter medication, herbal/nutraceutical preparation, within 7 days prior to enrollment.
5. Administration of any potentially nephrotoxic drug within 14 days prior to enrollment.
6. Use of an investigational drug and/or treatment within 30 days prior to enrollment.
7. Use of illicit drugs within 6 months prior to screening and enrollment, based on history and a urine drug screen.
8. Infection with HIV, HBV or HCV.
9. History of abuse of alcohol or other substance (s) within 6 months prior to enrollment.
10. History or symptoms of cardiovascular disease, including but not limited to coronary artery disease, hypertension, congestive heart disease, cardiomyopathy, and cardiac conduction disorders.
11. History of clinically significant hypotension (including orthostatic), fainting, or lightheadedness.
12. History of gastrointestinal disease or impairment.
13. History of renal impairment or disorder.
14. History of liver disease or impairment.
15. History of cancer, except basal cell carcinoma.
16. History of pathologic bone fractures; history or risk of osteopenia
17. History of diabetes, metabolic disease, or autoimmune disease; history of immunodeficiency in healthy volunteers.
18. Acute illness or fever 38 C within 1 week prior to enrollment.
19. Supine blood pressure - systolic outside the range of 90-140 mmHg, or diastolic outside the range of 50-90 mmHg.
20. Resting heart rate > 100 or < 45 beats per minute.
21. Body Mass Index (BMI) >31 or <18, or body weight <50 kg for men and < 45 kg for women.
22. Whole blood donation within 56 days or plasma donation within 30 days prior to enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Adverse events (AEs), absolute values and changes over time of clinical chemistry including troponin, hematology, and urinalysis, vital signs (blood pressure (BP) and heart rate), electrocardiogram | dosing-28 days post-dose

SECONDARY OUTCOMES:
CMX157 PK parameters: AUC(0-∞), AUC(0-t), Cmax, C12, and C24 following single dose administration. | dosin - 28 days post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Flach, MD, Principal Investigator — Covance
Locations (1):
- Covance, Madison, Wisconsin, United States